CLINICAL TRIAL: NCT00120965
Title: AutoPulse Assisted Prehospital International Resuscitation Trial (ASPIRE)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMB recommended termination due to lower survival to discharge in primary population and worse discharge CPC scores in the treatment arm than control arm.
Sponsor: University of Washington (Other)
Collaborators: Revivant Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-9613-B 01
Record Dates: First submitted 2005-06-30; First posted 2005-07-19 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Cardiac Arrest
Keywords: Cardiac arrest; OOH-cardiac arrest; CPR; Chest compressions; Chest compression device
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Autopulse device
  Interventions: Device: AutoPulse
- 2 (Active Comparator): Manual CPR
  Interventions: Other: Manual CPR

INTERVENTIONS:
Device: AutoPulse — Standard device settings
  Arms: 1
Other: Manual CPR — Manual CPR
  Arms: 2

SUMMARY:
The AutoPulse Assisted Prehospital International Resuscitation (ASPIRE) Trial compares the efficacy of circulatory assist by manual chest compression versus an automated chest compression device (AutoPulse™) during the resuscitative attempt following out-of-hospital cardiac arrest.

DETAILED DESCRIPTION:
Extensive early experience yielded no reliably validated instances of out-of-hospital arrest associated with tachyarrhythmia being resuscitated without successful defibrillatory shock. This together with the increasing availability of automated external defibrillators (AEDs), at increasingly attractive prices, led, in the past decade, to a strong emphasis on early defibrillation. This emphasis may have inadvertently resulted in a decreased emphasis on cardiopulmonary resuscitative techniques, particularly in light of publications decrying the uniformly poor quality of CPR performed by laymen, medical professionals, and even EMS personnel. However, recent research strongly suggests that assisted reperfusion prior to defibrillation may actually significantly improve survival rates. These reports, based on clinical studies, have received substantial confirmation from carefully controlled laboratory studies, particularly in pigs.

If assisted reperfusion prior to defibrillation (and subsequent to failed shock) is important, it is reasonable to suppose that the benefit is related to quality of chest compressions. Observations of resuscitative efforts in the field indicate that maintaining compressions is one of the more difficult tasks, for a variety of reasons. Observations in the laboratory with trained paramedics show that the depth of compression and the compression rate diminish rapidly with time from the onset of CPR, without the participant being aware that his/her effort is actually diminished.

The desire to provide consistent and quality compressions has led to the development of a mechanical compression assist device called the AutoPulse. It is a self-contained, portable chest compression device that is rapidly field deployable.

ELIGIBILITY:
Inclusion Criteria:

* All persons with out-of-hospital cardiac arrest who are attended by a vehicle involved in the randomization process and who are treated by the emergency medical service (EMS).

Exclusion Criteria:

* Persons under the age of 18
* Victims with traumatic arrest
* Less than the legal age of consent
* Resuscitation attempt discontinued because of do not resuscitate (DNR) orders or on request of authorized decision-maker
* Wards of the state, including prisoners
* Chest or abdominal surgery within 6 weeks
* Site specific exclusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1837 (Actual)
Dates: Start 2004-06; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Hospital admission defined as being alive four hours after the call for assistance to the emergency dispatch center.

SECONDARY OUTCOMES:
ROSC (a pulse in any vessel) at any time
ROSC at arrival to emergency department
Admittance to the hospital
Discharge from the hospital
CPC score at discharge from the hospital
Survival at 3 months post hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Alfred P. Hallstrom, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Clinical Trial Center, Seattle, Washington, United States

REFERENCES:
- [Result] Hallstrom A, Rea TD, Sayre MR, Christenson J, Anton AR, Mosesso VN Jr, Van Ottingham L, Olsufka M, Pennington S, White LJ, Yahn S, Husar J, Morris MF, Cobb LA. Manual chest compression vs use of an automated chest compression device during resuscitation following out-of-hospital cardiac arrest: a randomized trial. JAMA. 2006 Jun 14;295(22):2620-8. doi: 10.1001/jama.295.22.2620. PMID 16772625
- [Derived] Paradis NA, Young G, Lemeshow S, Brewer JE, Halperin HR. Inhomogeneity and temporal effects in AutoPulse Assisted Prehospital International Resuscitation--an exception from consent trial terminated early. Am J Emerg Med. 2010 May;28(4):391-8. doi: 10.1016/j.ajem.2010.02.002. PMID 20466215